CLINICAL TRIAL: NCT02211235
Title: Characterization of Glucose Variability by Continuous Glucose Monitoring in Non-diabetic Youth With and Without Cystic Fibrosis
Brief Title: Glycemic Monitoring in Cystic Fibrosis
Acronym: GEM
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-0960; UL1TR001082 (NIH)
Record Dates: First submitted 2014-07-29; First posted 2014-08-07 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Healthy Controls; Diabetes; Cystic Fibrosis Related Diabetes (CFRD); CFRD
MeSH Terms: conditions — Cystic Fibrosis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Alternative markers of glycemia, including fructosamine, glycated albumin, and 1,5-anhydroglucitol, Oral Glucose Tolerance Test (OGTT) derived markers of insulin secretion and insulin sensitivity
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Current guidelines on the diagnoses and management of cystic fibrosis (CF) related diabetes recommend treatment for diabetes based on diagnostic criteria derived from adults with type 2 diabetes. Increasing evidence supports treating early glucose abnormalities in cystic fibrosis patients to target CF specific outcomes, including lung function and nutrition (BMI-Body Mass Index). However, the criteria and timing of when to start insulin therapy in the 'prediabetic' state are unclear. A more accurate characterization of blood sugar variability in youth with and without CF will help the investigators better interpret continuous glucose monitor (CGM) findings in patients with CF prediabetes and diabetes and more accurately identify those individuals at greatest risk for disease progression.

ELIGIBILITY:
Inclusion Criteria:

Healthy controls (n=45) -

1. Age 10-25 years
2. BMI <85th percentile
3. Baseline health at enrollment

CF controls (n=45) -

1. Age 10-25 years
2. Diagnosis of cystic fibrosis (by newborn screen, sweat chloride testing, or genetic testing)
3. Baseline health at enrollment (no inclusion/exclusion criteria for CF patients based on lung function, BMI, pancreatic insufficiency, or genotype)

CF prediabetes & CFRD (n=70)

1. Age 10-25 years
2. Diagnosis of cystic fibrosis (by newborn screen, sweat chloride testing, or genetic testing)
3. History of abnormal oral glucose tolerance testing (2h-glucose >140, fasting plasma glucose >100,1hr glucose >200)
4. If taking medication that affects glucose metabolism (ex. Insulin, insulin sensitizers, glucocorticoids, atypical antipsychotics), should be on a stable dose over the past 3 months

Exclusion Criteria:

Healthy controls -

1. Known diagnosis of diabetes or prediabetes (including type 1, type 2, MODY), abnormal oral glucose tolerance test (OGTT) (ie. fasting plasma glucose ≥100 or 2hr ≥140 mg/dl) or HbA1c ≥ 5.7%
2. BMI ≥85th percentile
3. Chronic disease that may affect glucose metabolism or use of medications affecting glucose metabolism in the past 3 months (ex. Insulin, insulin sensitizers, glucocorticoids, atypical antipsychotics)
4. Presence of type 1 diabetes auto-antibodies in any individuals with a first degree relative with type 1 diabetes (will only include first degree relatives if they have had previous negative auto-antibody screening performed as part of participation in other studies such as the Trial Net studies at the Barbara Davis Center)
5. Acute illness (ex. Asthma exacerbation, gastroenteritis, febrile illness)
6. Pregnancy

CF participants -

1. Diagnosis of type 1 diabetes, type 2 diabetes, or MODY
2. Varying doses of medication affecting glucose metabolism in the past 3 months
3. Pulmonary exacerbation associated with hospitalization, or systemic steroid requirement in the preceding 6 weeks
4. Pregnancy

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children and Adolescents ages 6-25, without diabetes. Out of 160 people, 45 will be healthy controls, 45 with Cystic Fibrosis (normal glucose tolerance), and 70 with Cystic Fibrosis-related diabetes or pre-diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2014-08; Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
The percentage of time spent > 140 mg/dl on CGM | 7 days
  Percentage of time above normal glucose cut-point.

SECONDARY OUTCOMES:
The percentage of time spent > 120 mg/dl on CGM | 7 days
  Measures of glucose variability on CGM
The percentage of time spent > 200 mg/dl on CGM | 7 days
  Measures of glucose variability on CGM
The percentage of time spent < 70 mg/dl on CGM | 7 days
  Measures of glucose variability on CGM
The percentage of time spent < 60 mg/dl on CGM | 7 days
  Measures of glucose variability on CGM
The number of excursions > 200mg/dl in 24 hours for one week | 7 days
  Measures of glucose variability including peak glucose, mean glucose and measures of glucose variability on CGM.

OTHER OUTCOMES:
Change in CGM variables and BMI | 3 years
  To analyze in youth with CF the relationship between CGM variables and BMI Primary outcome: Change in BMI z-score collected at routine clinical visits over the preceding three years
Change in CGM variables and lung function | 3 years
  To analyze in youth with CF the relationship between CGM variables and lung function change in the preceding three years Secondary outcome: Change in forced expiratory volume at one second (FEV1) and forced vital capacity (FVC) measures collected at routine clinical visits over the preceding three years
Characterize the relationships between markers of glycemia | 3 days
  To characterize the relationships between alternative markers of glycemia (fructosamine, glycated albumin, and 1,5-anhydroglucitol) and CGM variables in non-diabetic CF youth and healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Christine L Chan, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Derived] Chan CL, Pyle L, Vigers T, Zeitler PS, Nadeau KJ. The Relationship Between Continuous Glucose Monitoring and OGTT in Youth and Young Adults With Cystic Fibrosis. J Clin Endocrinol Metab. 2022 Jan 18;107(2):e548-e560. doi: 10.1210/clinem/dgab692. PMID 34537845
- [Derived] Tommerdahl KL, Brinton JT, Vigers T, Cree-Green M, Zeitler PS, Nadeau KJ, Chan CL. Delayed glucose peak and elevated 1-hour glucose on the oral glucose tolerance test identify youth with cystic fibrosis with lower oral disposition index. J Cyst Fibros. 2021 Mar;20(2):339-345. doi: 10.1016/j.jcf.2020.08.020. Epub 2020 Sep 11. PMID 32928701
- [Derived] Chan CL, Hope E, Thurston J, Vigers T, Pyle L, Zeitler PS, Nadeau KJ. Hemoglobin A1c Accurately Predicts Continuous Glucose Monitoring-Derived Average Glucose in Youth and Young Adults With Cystic Fibrosis. Diabetes Care. 2018 Jul;41(7):1406-1413. doi: 10.2337/dc17-2419. Epub 2018 Apr 19. PMID 29674323